CLINICAL TRIAL: NCT00186771
Title: Transcranial Magnetic Stimulation Used to Treat Auditory Hallucinations in Schizophrenia
Brief Title: Magnetic Stimulation as a Treatment for Auditory Hallucinations in Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Dr. Gary Hasey, Director, TMS Laboratory, McMAster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMS-2363
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Schizophrenia
Keywords: Transcranial Magnetic Stimulation; Paired Pulse
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- True Transcranial Magnetic Stimulation (Active Comparator): True treatment with TMS over the temporoparietal cortex.
  Interventions: Device: Paired Pulse
- Sham Transcranial Magnetic Stimulation (Sham Comparator): Sham treatment with rTMS over the temporoparietal cortex.
  Interventions: Device: Paired Pulse

INTERVENTIONS:
Device: Paired Pulse — True treatment with rTMS over the temporoparietal cortex.
  Other Names: TMS
  Arms: True Transcranial Magnetic Stimulation
Device: Paired Pulse — Sham treatment with rTMS over the temporoparietal cortex.
  Other Names: TMS
  Arms: Sham Transcranial Magnetic Stimulation

SUMMARY:
Schizophrenia is a chronic, severe, and disabling brain disease. Auditory hallucinations are the most frequent symptoms with an incident of 50% to 70% in patients.

Transcranial Magnetic Stimulation (TMS) can significantly reduce symptoms of schizophrenia. TMS is capable of inducing changes in the electrical activities of the brain in humans.

The purpose of this trial is to study the use of TMS to decrease auditory hallucinations in schizophrenia.

DETAILED DESCRIPTION:
We hypothesize that: True treatment with rTMS will have significant decrease in auditory hallucinations versus sham treatment over the temporoparietal cortex.

FMRI will highlight areas of activation with auditory hallucinations distinct from the area identified by Hoffman's scalp based method.

Cortical inhibition as measured by paired pulse TMS will be increased after true TMS but not sham TMS.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia
* Auditory hallucinations occuring more than 5 times per day
* Adequate (6 weeks) trial of antipsychotic medication
* Including at least 1 atypical antipsychotic medication
* Medication stable for 4 weeks prior to commencement of the study
* Competent to consent

Exclusion Criteria:

* history of seizure disorder in patient or first degree relative
* recent head injury
* Acute suicidality
* Alcohol or substance abuse
* Implanted pacemaker or metal in head or neck
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2004-11; Primary Completion 2012-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Hoffman Auditory Hallucination Scale | weekly
  A series of 7 questions to identify the intensity and severity of the hallucinations

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale for Schizophrenia (PANSS) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hasey, MD, Principal Investigator — St. Joseph's Health Care London
Locations (1):
- St. Joseph's Healthcare, rTMS Laboratory, 100 West Fifth Street, Hamilton, Ontario, Canada